CLINICAL TRIAL: NCT04878354
Title: Efficacy and Safety of the SQ Tree Sublingual Immunotherapy Tablet in Children and Adolescents With Moderate to Severe Allergic Rhinitis and/or Conjunctivitis Induced by Pollen From Birch and Trees Belonging to the Birch Homologous Group
Brief Title: A Study in Children and Adolescents With Birch Pollen-induced Rhinoconjunctivitis
Acronym: TreeTop
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TT-06; 2020-004372-17 (EudraCT Number)
Record Dates: First submitted 2021-03-24; First posted 2021-05-07 (Actual); Results first posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Allergy
Keywords: Allergic rhinoconjunctivitis; Children; Adolescents; Birch
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Gelatine (fish source), mannitol and sodium hydroxide
  Interventions: Drug: Placebo SLIT-tablet
- Intervention/treatment (Experimental): Sublingual allergy immunotherapy tablet, for daily administration SQ tree SLIT-tablet
  Interventions: Drug: Tree SLIT-tablet

INTERVENTIONS:
Drug: Tree SLIT-tablet — Sublingual allergy immunotherapy tablets
  Arms: Intervention/treatment
Drug: Placebo SLIT-tablet — Placebo
  Arms: Placebo

SUMMARY:
This is a clinical study in children and adolescents (5-17 years) with allergy to pollen from birch (or related trees). It compares the tree SLIT-tablet with placebo in relieving rhinoconjunctivitis symptoms during the birch/tree pollen season based on the average allergic rhinoconjunctivitis daily total combined score.

The study will also collect health-related quality of life information in the groups treated with the tree SLIT-tablet or with placebo during the pollen season.

The trial medication used is already approved to treat allergic rhinitis caused by birch/tree pollen in adults in several countries?.

DETAILED DESCRIPTION:
This is a phase III, parallel-group, double-blind, placebo-controlled study to evaluate efficacy and safety of the tree SLIT-tablet in children and adolescents (5-17 years) who have rhinoconjunctivitis (with or without asthma) induced by pollen from birch trees or by trees belonging to the birch homologous group. Approximately 1000 children and adolescents will be enrolled in the trial and will receive either the tree SLIT-tablet or placebo.

The trial consists of 3 periods: a screening period, a treatment period, which includes pre-seasonal and co seasonal treatment, and a follow-up period. The duration is up to 13 months for each participant.

The trial is conducted in several European countries and in Canada.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of any race/ethnicity aged ≥4 to <18 years on the day informed consent is obtained from the parent/caregiver; the subject must be ≥5 to <18 years old at the randomisation visit
* A documented , physician diagnosed, clinically relevant history of moderate to severe AR/C induced by birch pollen (with or without asthma) despite having received treatment with symptom-relieving medication during at least 1 previous tree pollen season for ages 4 through 6 years at screening or at least 2 previous tree pollen seasons for ages 7 through 17 years at screening
* Positive skin prick test (SPT) to Betula verrucosa at screening
* Positive specific IgE to Bet v at screening
* Presence of 1 or more of the following Allergic Rhinitis Impact on Asthma (ARIA) quality of life items due to AR/C during the previous BPS:

  1. Sleep disturbance
  2. Impairment of daily activities, leisure and/or sport
  3. Impairment of school or work
  4. Troublesome symptoms

Exclusion Criteria:

* A clinically relevant history of symptomatic seasonal AR/C caused by an allergen source, other than tree pollen from the birch homologous group, with a season overlapping the TPS
* A clinically relevant history of symptomatic perennial AR/C caused by an allergen source such as animal hair and dander to which the subject is exposed during the TPS
* Any clinical deterioration of asthma (i.e. asthma exacerbation) that resulted in emergency treatment, hospitalisation or treatment with systemic corticosteroids within 3 months prior to randomisation
* Reduced lung function at randomisation defined as forced expiratory volume in 1 second (FEV1) <70% of predicted value. For subjects with asthma, this is assessed on subject's usual asthma medication following at least a 6-hour wash-out of SABA. This criterion does not need to be fulfilled if the subject is <7 years old, cannot perform reproducible FEV1 manoeuvres despite coaching and is not considered as having a diagnosis of asthma
* Ongoing treatment with any allergy immunotherapy product
* Severe chronic oral inflammation
* A diagnosis of eosinophilic oesophagitis
* A relevant history of systemic allergic reaction e.g. anaphylaxis with cardiorespiratory symptoms, generalised urticaria or severe facial angioedema that in the opinion of the investigator may constitute an increased safety concern
* Immunosuppressive treatment (ATC code L04 or L01) within 3 months prior to the screening visit

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 952 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monika Gappa, Prof. MD, Principal Investigator — Evangelisches Krankenhaus Düsseldorf
Locations (79):
- Austria (2):
  - Allergy Center Vienna West, Vienna
  - Medical University of Vienna, Vienna
- Belgium (3):
  - Practice Dr Jean-Benoit Martinot, Erpent, Namur
  - Universitair Ziekenhuis Gent, Ghent, Oost-Vlandeeren
  - UZ Leuven, Leuven, Vlaams Brabant
- Canada (2):
  - CHU Sainte-Justine, Montreal, Quebec
  - Clinique specialisee en allergie de la capitale, Québec
- Denmark (3):
  - Aarhus Universitetshospital, Astma, Allergi- og Lungeklinikken for Born, Aarhus
  - Astma, Allergi- og Lungeklinik, Copenhagen
  - Gentofte Hospital Allergy Clinic, Hellerup
- Germany (17):
  - Kinder- u. Jugendmedizin, Heidelberg, Baden-Wurttemberg
  - Gemeinschaftspraxis für Kinder und Jugendmedizin, Mannheim, Baden-Wurttemberg
  - Klinikum rechts der Isar der TUM, Munich, Bavaria
  - Universitätsklinikum Gießen und Marburg GmbH - Klinik für Hals-, Nasen- und Ohrenheilkunde Sektion Rhinologie und Allergologie, Marburg, Hesse
  - KliFOs - Klinische Forschung Osnabrück, Osnabrück, Lower Saxony
  - Evangelisches Krankenhaus Düsseldorf - Klinik für Kinder- und Jugendmedizin, Düsseldorf, North Rhine-Westphalia
  - ENT Research GmbH, Essen, North Rhine-Westphalia
  - Kinder- und Jugendärzte, Hürth, North Rhine-Westphalia
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - Praxis Dr.J. Funck, Neuss, North Rhine-Westphalia
  - Praxis Dr. med. Karsten Jünger, Herxheim, Rhineland-Palatinate
  - Universitätsmedizin der JGU, Mainz, Rhineland-Palatinate
  - Kinderarztpraxis Dr. med. Siegfried Simmet und Simon Traub, Schweigen-Rechtenbach, Rhineland-Palatinate
  - Praxis Dr. Yury Yarin, Dresden, Saxony
  - HNO Praxis Dr. Uta Thieme, Duisburg
  - Hautarztpraxis Dr. med. Daniela Kasche, Hamburg
  - HNO-Praxis am Neckar, Heidelberg
- Hungary (5):
  - Aranyklinika Kft, Szeged, Csongrád megye
  - Svábhegy Plusz Kft, Budapest
  - Semmelweis Egyetem, Budapest
  - Heim Pál Gyermekkórház, Budapest
  - Kispesti Egeszsegugyi Intezet, Budapest
- Lithuania (9):
  - JSC Ausros Medicinos Centras, Kaunas, Kaunas County
  - "CD8 Klinika" JSC, Kaunas, Kaunas County
  - "Medicum centrum" JSC, Tauragė, Tauragė County
  - "Seimos gydytojas" JSC, Vilnius, Vilnius County
  - "Inlita" JSC Santara CTC, Vilnius, Vilnius County
  - Allergy clinic "Perspektyvos" JSC, Vilnius, Vilnius County
  - Hospital of University of Health Sciences Kauno Klinikos, Kaunas
  - Alerginiu susirgimu diagnostikos ir gydymo centras, Vilnius
  - "Center of Innovative Allergology" JSC, Vilnius
- Netherlands (2):
  - Medisch Spectrum Twente, Enschede, Overijssel
  - Erasmus MC - Sophia Childrens Hospital, Rotterdam, South Holland
- Poland (23):
  - Centrum Medyczne PRATIA Bydgoszcz, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Centrum Medyczne ALL-MED, Krakow, Lesser Poland Voivodeship
  - Centrum Medyczne PROMED, Krakow, Lesser Poland Voivodeship
  - Malopolskie Centrum Alergologii, Krakow, Lesser Poland Voivodeship
  - ALERGO-MED Spolka z o.o., Tarnów, Lesser Poland Voivodeship
  - Centrum Alergologii Specjalistyczna Przychodnia Alergologiczna, Lublin, Lublin Voivodeship
  - NZOZ E-Vita, Bialystok, Podlaskie Voivodeship
  - Specjalist. Praktyka Lek. dr n.med. Joanna Orlicz-Widawska, Katowice, Silesian Voivodeship
  - Niepubliczny Zaklad Opieki Zdrowotnej "ALERGOLOGIA", Poradnia Alergologiczna, Szczecin, West Pomeranian Voivodeship
  - Centrum Medyczne Pratia Czestochowa, Częstochowa
  - Indywidualna Specjalistyczna Praktyka Lekarska lek. med. Elzbieta Matusz, Gryfice
  - ETG Kielce, Kielce
  - Centrum Medyczne Plejady, Krakow
  - SPZOZ Uniwersytecki Szpital Kliniczny nr 1 im. N.Barlickiego, Lodz
  - WWCOiT im. M. Kopernika w Lodzi, Osrodek Pediatryczny im. dr J.Korczaka, Lodz
  - Centrum Alergologii Prof. K. Buczyłko Spółka z o.o., Lodz
  - Alergotest s.c. Specjalistyczne Centrum Medyczne, Lublin
  - Gabinet Lekarski Pediatryczno-Alergologiczny Zenon Bukowczan, Sucha Beskidzka
  - "All-Med" Specjalistyczna Opieka Medyczna, Wroclaw
  - Michal Bogacki DOBROSTAN, Wroclaw
  - Niepubliczny Zaklad Opieki Zdrowotnej Centrum Uslug Medycznych "PROXIMUM" Sp. z o.o., Wroclaw
  - ETG Skierniewice, Skierniewice, Łódź Voivodeship
  - NSZOZ Puls - Med Anna Bogusz, Agnieszka Musielak Sp.J., Skarżysko-Kamienna, Świętokrzyskie Voivodeship
- Russia (5):
  - LLC "Olla-Med", Moscow, Moscow
  - NRPC Pediatric Hematology, Oncology, Immunology n.a. Dmitriya Rogacheva - Multispecialty, Moscow, Moscow
  - FGBU "Scientific center of children health" of RAMS, Moscow, Moscow
  - Public Enterprise State Scient, Moscow
  - FGBUN" Federal Research Center for Nutrition and Biotechnology ", Moskva
- Slovakia (8):
  - ALERGO H2B s.r.o., Komárno, Nitra Region
  - DANIMED, spol. s.r.o., Levice
  - Univerzitna Nemocnica Martin, Martin
  - MedKol, s.r.o., Nové Zámky
  - EMED s.r.o., Prešov
  - Zoll-Med s.r.o., Ambulancia klinickej imunologie a alergologie, Rimavská Sobota
  - Ambulancia klinickej imunologie a alergologie, Šurany
  - SIMIDA s.r.o., Vráble

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 952 participants were randomized and treated. Participants were recruited from 80 sites in 11 countries (Austria, Belgium, Canada, Denmark, Germany, Hungary, Lithuania, Netherlands, Poland, Russia and Slovakia). First participant first visit: 08-Apr-2021. Last participant last visit/contact: 31-Jul-2023.
Pre-assignment Details: * Male or female aged ≥5 to <18 years at randomization
  * Documented, clinically relevant history of moderate to severe allergic rhinitis and/or conjunctivitis (AR/C) induced by birch pollen (with or without asthma) despite treatment with symptom-relieving medication
  * Positive skin prick test (SPT) and IgE against Betula verrucosa
  * Presence of at least 1 Allergic Rhinitis Impact on Asthma (ARIA) quality of life item due to AR/C during the previous birch pollen season (BPS)
Groups:
- Placebo SLIT-tablet: Participants received 1 placebo sublingual immunotherapy (SLIT)-tablet daily plus rhinoconjunctivitis rescue medication as needed.
- Tree SLIT-tablet: Participants received 1 tree sublingual immunotherapy (SLIT)-tablet, 12 SQ-Bet dose daily plus rhinoconjunctivitis rescue medication as needed.
Period: Overall Study
Arm/Group | Placebo SLIT-tablet | Tree SLIT-tablet
Started (Randomized and treated) | 479 | 473
Completed Trial | 458 | 456
Full Analysis Set (Full analysis set, defined as all randomized participants. Participants were analyzed as randomized i.e., according to their randomized assignment of treatment) | 479 | 473
Safety Analysis Set (Safety analysis set definded as all randomized participants who received at least one dose of IMP. Participants were analyzed as treated i.e., according to treatment they actually received) | 479 | 473
Subgroup Analysis Set (Participants in a random subset sample stratified by treatment group and age group for cohort 1. The subgroup is used for immunology assessment) | 132 | 119
Completed (Completed IMP) | 454 | 443
Not Completed | 25 | 30
Not completed — Adverse Event | 4 | 13
Not completed — Withdrawal by Subject | 14 | 12
Not completed — Lost to Follow-up | 4 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Reason stated as "other" in CRF | 2 | 3

BASELINE CHARACTERISTICS:
Population: All randomized and treated participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo SLIT-tablet | Tree SLIT-tablet | Total
Number analyzed (Participants) | 479 | 473 | 952
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 479 | 473 | 952
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.2 (3.5) | 10.4 (3.5) | 10.3 (3.5)
Age, Customized [Count of Participants; unit: Participants] — Participants aged ≥5 to <18 years
  Participants
    Age by group: 5-11 years | 300 | 297 | 597
    Age by group: 12-17 years | 179 | 176 | 355
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 194 | 185 | 379
  Male | 285 | 288 | 573
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 471 | 463 | 934
  Unknown or Not Reported | 3 | 7 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4 | 1 | 5
  White | 473 | 468 | 941
  Black or African American | 0 | 1 | 1
  Multiple | 2 | 2 | 4
  Other | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 42 | 45 | 87
  Austria | 4 | 6 | 10
  Netherlands | 2 | 0 | 2
  Belgium | 3 | 4 | 7
  Hungary | 24 | 21 | 45
  Denmark | 10 | 8 | 18
  Poland | 225 | 221 | 446
  Slovakia | 40 | 39 | 79
  Lithuania | 46 | 46 | 92
  Germany | 44 | 45 | 89
  Russia | 39 | 38 | 77
Allergic condition caused by birch [Number; unit: participants]
  Allergic conjunctivitis | 4 | 2 | 6
  Allergic rhinitis | 122 | 125 | 247
  Allergic rhinoconjunctivitis | 353 | 346 | 699
  Asthma | 125 | 126 | 251

OUTCOME MEASURES:

1. Primary Outcome: Average Total Combined Score (TCS) During the Birch Pollen Season (BPS)
Description: The primary endpoint of the trial was the average allergic rhinitis and/or conjunctivitis TCS during the BPS. The average TCS evaluates the treatment effect based on reduction in daily rhinoconjunctivitis symptoms and medication use (on a scale of 0-38). Higher scores indicate more severe symptoms and/or more medication use. The endpoint is calculated as the average score of all reported daily values during the BPS. The primary estimand for the endpoint was the trial product estimand. The trial product estimand assesses the anticipated effect of the tree SLIT-tablet if it is taken as instructed.
Time Frame: During the BPS (mean duration of approximately 3-4 weeks)
Population: Participants in the full analysis set with observations
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo SLIT-tablet | Tree SLIT-tablet
Number analyzed (Participants) | 457 | 444
score on a scale | 5.88 (0.33) | 4.60 (0.29)
Statistical Analysis 1: Comparison: Placebo SLIT-tablet vs Tree SLIT-tablet; Multiple imputation was used to impute missing data under the hypothetical strategy. The square root transformed endpoint was analysed in a linear mixed effects (LME) model with treatment, cohort, and age group as fixed effects, and pollen station within cohort as a random effect with different residual errors specified for each treatment group. Back-transformation was used to estimate the absolute difference. Adjusted p-value; Test type: Superiority; p = 0.0004, Mixed Models Analysis; Mean Difference (Final Values) = 1.29, 95% CI 2-sided [0.58 to 2.00] — Placebo SLIT-tablet vs. tree SLIT-tablet

2. Secondary Outcome: Average Total Combined Score (TCS) During the Tree Pollen Season (TPS)
Description: Average TCS measured in the TPS. TPS includes hazel, alder, birch and oak pollen seasons. The average TCS evaluates the treatment effect based on reduction in daily rhinoconjunctivitis symptoms and medication use (on a scale of 0-38). Higher scores indicate more severe symptoms and/or more medication use. The endpoint is calculated as the average score of all reported daily values during the TPS. The primary estimand for the endpoint was the trial product estimand. The trial product estimand assesses the anticipated effect of the tree SLIT-tablet if it is taken as instructed.
Time Frame: During the TPS (mean duration of approximately 11 weeks)
Population: Participants in the full analysis set with observations
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo SLIT-tablet | Tree SLIT-tablet
Number analyzed (Participants) | 461 | 448
score on a scale | 4.51 (0.25) | 3.66 (0.22)
Statistical Analysis 1: Comparison: Placebo SLIT-tablet vs Tree SLIT-tablet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0010, Mixed Models Analysis; Mean Difference (Final Values) = 0.85, 95% CI 2-sided [0.34 to 1.35] — Placebo SLIT-tablet vs. tree SLIT-tablet

3. Secondary Outcome: Average Daily Symptoms Score (DSS) During the Birch Pollen Season (BPS)
Description: Average rhinoconjunctivitis DSS during the BPS evaluates the treatment effect based on the reduction in daily rhinoconjunctivitis symptoms (on a scale of 0 to 18). Higher scores indicate more severe symptoms. The endpoint is calculated as the average score of all reported daily values during the BPS. The primary estimand for the endpoint was the trial product estimand. The trial product estimand assesses the anticipated effect of the tree SLIT-tablet if it is taken as instructed.
Time Frame: During the BPS (mean duration of approximately 3-4 weeks)
Population: Participants in the full analysis set with observations
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo SLIT-tablet | Tree SLIT-tablet
Number analyzed (Participants) | 457 | 444
score on a scale | 2.75 (0.16) | 2.39 (0.15)
Statistical Analysis 1: Comparison: Placebo SLIT-tablet vs Tree SLIT-tablet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0354, Mixed Models Analysis; Mean Difference (Final Values) = 0.37, 95% CI 2-sided [0.03 to 0.71] — Placebo SLIT-tablet vs. tree SLIT-tablet

4. Secondary Outcome: Average Daily Symptoms Score (DSS) During the Tree Pollen Season (TPS)
Description: Average rhinoconjunctivitis DSS during the TPS evaluates the treatment effect based on the reduction in daily rhinoconjunctivitis symptoms (on a scale of 0 to 18). TPS includes hazel, alder, birch and oak pollen seasons. Higher scores indicate more severe symptoms. The endpoint is calculated as the average score of all reported daily values during the TPS. The primary estimand for the endpoint was the trial product estimand. The trial product estimand assesses the anticipated effect of the tree SLIT-tablet if it is taken as instructed.
Time Frame: During the TPS (mean duration of approximately 11 weeks).
Population: Participants in the full analysis set with observations
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo SLIT-tablet | Tree SLIT-tablet
Number analyzed (Participants) | 461 | 448
score on a scale | 2.28 (0.14) | 2.04 (0.13)
Statistical Analysis 1: Comparison: Placebo SLIT-tablet vs Tree SLIT-tablet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0734, Mixed Models Analysis; Mean Difference (Final Values) = 0.24, 95% CI 2-sided [-0.02 to 0.50] — Placebo SLIT-tablet vs. tree SLIT-tablet

5. Secondary Outcome: Average Daily Medication Score (DMS) During the Birch Pollen Season (BPS)
Description: Average rhinoconjunctivitis DMS during the BPS evaluates the treatment effect based on the reduction in daily rhinoconjunctivitis medication use (on a scale of 0 to 20). Higher scores indicate more medication use. The endpoint is calculated as the average score of all reported daily values during the BPS. The primary estimand for the endpoint was the trial product estimand. The trial product estimand assesses the anticipated effect of the tree SLIT-tablet if it is taken as instructed.
Time Frame: During the BPS (mean duration of approximately 3-4 weeks)
Population: Participants in the full analysis set with observations.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo SLIT-tablet | Tree SLIT-tablet
Number analyzed (Participants) | 457 | 444
score on a scale | 2.42 (0.23) | 1.55 (0.18)
Statistical Analysis 1: Comparison: Placebo SLIT-tablet vs Tree SLIT-tablet; Multiple imputation was used to impute missing data under the hypothetical strategy. The square root transformed endpoint was analysed in a linear mixed effects (LME) model with treatment, cohort, and age group as fixed effects, and pollen station within cohort as a random effect with different residual errors specified for each treatment group. Back-transformation was used to estimate the absolute difference. Observed p-value; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.86, 95% CI 2-sided [0.45 to 1.28] — Placebo SLIT-tablet vs. tree SLIT-tablet

6. Secondary Outcome: Average Daily Medication Score (DMS) During the Tree Pollen Season (TPS)
Description: Average rhinoconjunctivitis DMS during the TPS evaluates the treatment effect based on the reduction in daily rhinoconjunctivitis medication use (on a scale of 0 to 20). TPS includes hazel, alder, birch and oak pollen seasons. Higher scores indicate more medication use. The endpoint is calculated as the average score of all reported daily values during the TPS. The primary estimand for the endpoint was the trial product estimand. The trial product estimand assesses the anticipated effect of the tree SLIT-tablet if it is taken as instructed.
Time Frame: During the TPS (mean duration of approximately 11 weeks)
Population: Participants in the full analysis set with observations
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo SLIT-tablet | Tree SLIT-tablet
Number analyzed (Participants) | 461 | 448
score on a scale | 1.72 (0.16) | 1.18 (0.13)
Statistical Analysis 1: Comparison: Placebo SLIT-tablet vs Tree SLIT-tablet; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.0002, Mixed Models Analysis; Mean Difference (Final Values) = 0.54, 95% CI 2-sided [0.26 to 0.82] — Placebo SLIT-tablet vs. tree SLIT-tablet

7. Secondary Outcome: Average Total Combined Score (TCS) During the Alder Hazel Pollen Season (AHPS)
Description: Average TCS during the AHPS evaluates the treatment effect based on reduction in daily rhinoconjunctivitis symptoms and medication use (on a scale of 0-38). Higher scores indicate more severe symptoms and/or more medication use. The endpoint is calculated as the average score of all reported daily values during the AHPS. The primary estimand for the endpoint was the trial product estimand. The trial product estimand assesses the anticipated effect of the tree SLIT-tablet if it is taken as instructed.
Time Frame: During the AHPS (mean duration of approximately 6-7 weeks)
Population: Participants in the full analysis set with observations
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo SLIT-tablet | Tree SLIT-tablet
Number analyzed (Participants) | 442 | 426
score on a scale | 2.83 (0.22) | 2.51 (0.21)
Statistical Analysis 1: Comparison: Placebo SLIT-tablet vs Tree SLIT-tablet; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.1516, Mixed Models Analysis; Mean Difference (Final Values) = 0.32, 95% CI 2-sided [-0.11 to 0.76] — Placebo SLIT-tablet vs. tree SLIT-tablet

8. Secondary Outcome: Average Daily Symptoms Score (DSS) During the Alder Hazel Pollen Season (AHPS)
Description: Average rhinoconjunctivitis DSS during the AHPS evaluates the treatment effect based on the reduction in daily rhinoconjunctivitis symptoms (on a scale of 0 to 18). Higher scores indicate more severe symptoms. The endpoint is calculated as the average score of all reported daily values during the AHPS. The primary estimand for the endpoint was the trial product estimand. The trial product estimand assesses the anticipated effect of the tree SLIT-tablet if it is taken as instructed.
Time Frame: During the AHPS (mean duration of approximately 6-7 weeks)
Population: Participants in the full analysis set with observations
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo SLIT-tablet | Tree SLIT-tablet
Number analyzed (Participants) | 442 | 426
score on a scale | 1.57 (0.12) | 1.56 (0.13)
Statistical Analysis 1: Comparison: Placebo SLIT-tablet vs Tree SLIT-tablet; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.9709, Mixed Models Analysis; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.24 to 0.25] — Placebo SLIT-tablet vs. tree SLIT-tablet

9. Secondary Outcome: Average Daily Medication Score (DMS) During the Alder Hazel Pollen Season (AHPS)
Description: Average rhinoconjunctivitis DMS during the AHPS evaluates the treatment effect based on the reduction in daily rhinoconjunctivitis medication use (on a scale of 0 to 20). Higher scores indicate more medication use. The endpoint is calculated as the average score of all reported daily values during the AHPS. The primary estimand for the endpoint was the trial product estimand. The trial product estimand assesses the anticipated effect of the tree SLIT-tablet if it is taken as instructed.
Time Frame: During the AHPS (mean duration of approximately 6-7 weeks)
Population: Participants in the full analysis set with observations
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo SLIT-tablet | Tree SLIT-tablet
Number analyzed (Participants) | 442 | 426
score on a scale | 0.80 (0.11) | 0.59 (0.09)
Statistical Analysis 1: Comparison: Placebo SLIT-tablet vs Tree SLIT-tablet; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.0499, Mixed Models Analysis; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [0.00 to 0.41] — Placebo SLIT-tablet vs. tree SLIT-tablet

10. Secondary Outcome: Average Total Combined Score (TCS) During the Oak Pollen Season (OPS)
Description: Average TCS measured in the OPS evaluates the treatment effect based on reduction in daily rhinoconjunctivitis symptoms and medication use (on a scale of 0-38). Higher scores indicate more severe symptoms and/or more medication use. The endpoint is calculated as the average score of all reported daily values during the OPS. The primary estimand for the endpoint was the trial product estimand. The trial product estimand assesses the anticipated effect of the tree SLIT-tablet if it is taken as instructed.
Time Frame: During the OPS (mean duration of approximately 3 weeks)
Population: Participants in the full analysis set with observations
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo SLIT-tablet | Tree SLIT-tablet
Number analyzed (Participants) | 442 | 432
score on a scale | 5.67 (0.36) | 4.22 (0.31)
Statistical Analysis 1: Comparison: Placebo SLIT-tablet vs Tree SLIT-tablet; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Median Difference (Final Values) = 1.45, 95% CI 2-sided [0.73 to 2.18] — Placebo SLIT-tablet vs. tree SLIT-tablet

11. Secondary Outcome: Average Daily Symptoms Score (DSS) During the Oak Pollen Season (OPS)
Description: Average rhinoconjunctivitis DSS during the OPS evaluates the treatment effect based on the reduction in daily rhinoconjunctivitis symptoms (on a scale of 0 to 18). Higher scores indicate more severe symptoms. The endpoint is calculated as the average score of all reported daily values during the OPS. The primary estimand for the endpoint was the trial product estimand. The trial product estimand assesses the anticipated effect of the tree SLIT-tablet if it is taken as instructed.
Time Frame: During the OPS (mean duration of approximately 3 weeks)
Population: Participants in the full analysis set with observations.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo SLIT-tablet | Tree SLIT-tablet
Number analyzed (Participants) | 442 | 432
score on a scale | 2.68 (0.16) | 2.20 (0.15)
Statistical Analysis 1: Comparison: Placebo SLIT-tablet vs Tree SLIT-tablet; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.0075, Mixed Models Analysis; Median Difference (Final Values) = 0.48, 95% CI 2-sided [0.13 to 0.83] — Placebo SLIT-tablet vs. tree SLIT-tablet

12. Secondary Outcome: Average Daily Medication Score (DMS) During the Oak Pollen Season (OPS)
Description: Average rhinoconjunctivitis DMS during the OPS evaluates the treatment effect based on the reduction in daily rhinoconjunctivitis medication use (on a scale of 0 to 20). Higher scores indicate more medication use. The endpoint is calculated as the average score of all reported daily values during the OPS. The primary estimand for the endpoint was the trial product estimand. The trial product estimand assesses the anticipated effect of the tree SLIT-tablet if it is taken as instructed.
Time Frame: During the OPS (mean duration of approximately 3 weeks)
Population: Participants in the full analysis set with observations
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo SLIT-tablet | Tree SLIT-tablet
Number analyzed (Participants) | 442 | 432
score on a scale | 2.18 (0.23) | 1.31 (0.18)
Statistical Analysis 1: Comparison: Placebo SLIT-tablet vs Tree SLIT-tablet; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Median Difference (Final Values) = 0.87, 95% CI 2-sided [0.44 to 1.29] — Placebo SLIT-tablet vs. tree SLIT-tablet

13. Secondary Outcome: Number of Severe Days During the Birch Pollen Season (BPS)
Description: The disease burden for participants was analyzed in terms of proportion of severe days.
  A severe day was a day with a daily symptom score (DSS) ≥6 and ≥2 moderate symptoms or 1 severe symptom. The DSS ranged from 0 to 18 and was the sum of the 6 allergic rhinoconjunctivitis symptom scores, each scored on a scale from 0 to 3 (0 = no symptoms, 1= mild symptoms, 2= moderate symptoms and 3 = severe symptoms).
  The proportion of severe days was the number of severe days divided by the number of days in the season.
Time Frame: During the BPS (mean duration of approximately 3-4 weeks)
Population: Participants in the full analysis set with observations
Measure: Number; unit: Proportion of severe days
Arm/Group | Placebo SLIT-tablet | Tree SLIT-tablet
Number analyzed (Participants) | 457 | 444
Proportion of severe days | 0.23 | 0.20
Statistical Analysis 1: Comparison: Placebo SLIT-tablet vs Tree SLIT-tablet; The odds of having a severe day was analysed using a generalised linear mixed model (GLMM) with a logit link function. The model includes proportion of severe days as the response variable and treatment, cohort, and age group as fixed effects and pollen station as random effect. Observed p-value; Test type: Superiority; p < 0.0001, Generalised linear mixed model (GLMM); Odds Ratio (OR) = 1.20, 95% CI 2-sided [1.10 to 1.32] — Odds ratio is (odds placebo SLIT-tablet / odds tree SLIT-tablet)

14. Secondary Outcome: Number of Severe Days During the Tree Pollen Season (TPS)
Description: as for outcome 13
Time Frame: During the TPS (mean duration of approximately 11 weeks)
Population: Participants in the full analysis set with observations.
Measure: Number; unit: Proportion of severe days
Arm/Group | Placebo SLIT-tablet | Tree SLIT-tablet
Number analyzed (Participants) | 461 | 448
Proportion of severe days | 0.11 | 0.11
Statistical Analysis 1: Comparison: Placebo SLIT-tablet vs Tree SLIT-tablet; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.9124, Generalised linear mixed model (GLMM); Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.93 to 1.08] — Odds ration is (odds placebo SLIT-tablet / odds tree SLIT-tablet)

15. Secondary Outcome: Number of Well Days During the Birch Pollen Season (BPS)
Description: A well day was defined as a day with no use of allergic rhinitis and/or conjunctivitis (AR/C) rescue medication (daily medication score =0) and daily symptom score ≤2.
  The proportion of well days was the number of well days divided by the number of days in the season.
Time Frame: During the BPS (mean duration of approximately 3-4 weeks)
Population: Participants in the full analysis set with observations
Measure: Number; unit: Proportion of well days
Arm/Group | Placebo SLIT-tablet | Tree SLIT-tablet
Number analyzed (Participants) | 457 | 444
Proportion of well days | 0.36 | 0.43
Statistical Analysis 1: Comparison: Placebo SLIT-tablet vs Tree SLIT-tablet; The odds of having a well day was analysed using a generalised linear mixed model (GLMM) with a logit link function. The model includes proportion of well days as the response variable and treatment, cohort, and age group as fixed effects and pollen station as random effect. Observed p-value; Test type: Superiority; p < 0.0001, Generalised linear fixed model (GLMM); Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.71 to 0.81] — Odds ratio is (odds placebo SLIT-tablet / odds tree SLIT-tablet)

16. Secondary Outcome: Number of Well Days During the Tree Pollen Season (TPS)
Description: as for outcome 15
Time Frame: During the TPS (mean duration of approximately 11 weeks)
Population: Participants in the full analysis set with observations.
Measure: Number; unit: Proportion of well days
Arm/Group | Placebo SLIT-tablet | Tree SLIT-tablet
Number analyzed (Participants) | 461 | 448
Proportion of well days | 0.50 | 0.53
Statistical Analysis 1: Comparison: Placebo SLIT-tablet vs Tree SLIT-tablet; [analysis description as in outcome 15, analysis 1]; Test type: Superiority; p < 0.0001, Generalised linear mixed model (GLMM); Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.85 to 0.93] — Odds ratio is (odds placebo SLIT-tablet / odds tree SLIT-tablet)

17. Secondary Outcome: Number of Symptom-free Days During the Birch Pollen Season (BPS)
Description: A a symptom-free day was defined as a day with no symptoms and with no use of rescue medication (Total Combined Score = 0). The proportion of symptom-free days was the number of symptom-free divided by the number of days in the season.
Time Frame: During the BPS (mean duration of approximately 3-4 weeks)
Population: Participants in the full analysis set with observations
Measure: Number; unit: Proportion of symptom-free days
Arm/Group | Placebo SLIT-tablet | Tree SLIT-tablet
Number analyzed (Participants) | 457 | 444
Proportion of symptom-free days | 0.24 | 0.29
Statistical Analysis 1: Comparison: Placebo SLIT-tablet vs Tree SLIT-tablet; The odds of having a symptom-free day was analysed using a generalised linear mixed model (GLMM) with a logit link function. The model includes proportion of symptom-free days as the response variable and treatment, cohort, and age group as fixed effects and pollen station as random effect. Observed p-value; Test type: Superiority; p < 0.0001, Generalised linear mixed model (GLMM); Odds Ratio (OR) = 0.78, 95% CI 2-sided [0.72 to 0.84] — Odds ratio is (odds placebo SLIT-tablet / odds tree SLIT-tablet)

18. Secondary Outcome: Number of Symptom-free Days During the Tree Pollen Season (TPS)
Description: as for outcome 17
Time Frame: During the TPS (mean duration of approximately 11 weeks)
Population: Participants in the full analysis set with observations
Measure: Number; unit: Proportion of symptom-free days
Arm/Group | Placebo SLIT-tablet | Tree SLIT-tablet
Number analyzed (Participants) | 461 | 448
Proportion of symptom-free days | 0.28 | 0.30
Statistical Analysis 1: Comparison: Placebo SLIT-tablet vs Tree SLIT-tablet; [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p = 0.0001, Generalised linear mixed model (GLMM); Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.86 to 0.95] — Odds ratio is (odds placebo SLIT-tablet / odds tree SLIT-tablet)

19. Secondary Outcome: Percentage of Patients Free of Symptoms and With no Use of Rescue Medication During the Birch Pollen Season (BPS)
Description: A symptom-free day was defined as a day with no symptoms and with no use of rescue medication, i.e. total combined score (TCS) =0. Thus, the endpoint was categorized as a binary variable with a subject being a responder if he/she had no symptoms and had not used rescue medication during the season
Time Frame: During the BPS (mean duration of approximately 3-4 weeks)
Population: Participants in the full analysis set with observations
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo SLIT-tablet | Tree SLIT-tablet
Number analyzed (Participants) | 479 | 473
Participants
  No season data | 19 | 18
  TCS=0 all days | 21 | 20
  TCS> 0 any day | 439 | 435

20. Secondary Outcome: Percentage of Patients Free of Symptoms and With no Use of Rescue Medication During the Tree Pollen Season (TPS)
Description: A symptom-free day was defined as a day with no symptoms and with no use of rescue medication, i.e. total combined score (TCS) = 0. Thus, the endpoint was categorized as a binary variable with a subject being a responder if he/she had no symptoms and had not used rescue medication during the tree pollen season.
Time Frame: During the TPS (mean duration of approximately 11 weeks)
Population: Participants in the full analysis set with observations
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo SLIT-tablet | Tree SLIT-tablet
Number analyzed (Participants) | 479 | 473
Participants
  No season data | 15 | 16
  TCS = 0 all days | 10 | 4
  TCS > 0 any day | 454 | 453

21. Secondary Outcome: Average Total Combined Score (TCS) (EAACI Scoring) During Birch Pollen Season (BPS)
Description: The TCS European Academy of Allergy and Clinical Immunology (EAACI) scoring was calculated using the medication score proposed by EAACI and was the sum of the DSS/6 and the daily EAACI medication score (DMSEAACI) (values 0,1,2), and thus ranged 0-5 with higher scores indicating more combined allergy symptoms and medication use. The primary estimand for the endpoint was the trial product estimand. The trial product estimand assesses the anticipated effect of the tree SLIT-tablet if it is taken as instructed.
Time Frame: During the BPS (mean duration of approximately 3-4 weeks)
Population: Participants in the full analysis set with observations
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo SLIT-tablet | Tree SLIT-tablet
Number analyzed (Participants) | 457 | 444
score on a scale | 0.95 (0.05) | 0.77 (0.05)
Statistical Analysis 1: Comparison: Placebo SLIT-tablet vs Tree SLIT-tablet; Multiple imputation was used to impute missing data under the hypothetical strategy. The square root transformed endpoint was analysed in an LME model with treatment, cohort, and age group as fixed effects, and pollen station within cohort as a random effect with different residual errors specified for each treatment group. Back-transformation was used to estimate the absolute difference. Observed p-value; Test type: Superiority; p = 0.0015, Mixed Models Analysis; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [0.07 to 0.29] — Placebo SLIT-tablet vs tree SLIT-tablet

22. Secondary Outcome: Average Total Combined Score (TCS) (EAACI Scoring) During Tree Pollen Season (TPS)
Description: as for outcome 21
Time Frame: During the TPS (mean duration of approximately 11 weeks).
Population: Participants in the full analysis set with observations
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo SLIT-tablet | Tree SLIT-tablet
Number analyzed (Participants) | 461 | 448
score on a scale | 0.74 (0.04) | 0.62 (0.04)
Statistical Analysis 1: Comparison: Placebo SLIT-tablet vs Tree SLIT-tablet; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.0032, Mixed Models Analysis; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [0.04 to 0.20] — Placebo SLIT-tablet vs tree SLIT-tablet

23. Secondary Outcome: Average Weekly Overall Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Score During the Birch Pollen Season (BPS) (12-17 Years Only)
Description: The RQLQ measured the rhinoconjunctivitis quality of life. The RQLQ (for participants 12-17 years only) comprised 28 items, each scored on a 7-point scale ranging 0-6, with higher scores indicating worse quality of life. The overall RQLQ score was the mean of the 28 item scores.
  The primary estimand for the endpoint was the trial product estimand. The trial product estimand assesses the anticipated effect of the tree SLIT-tablet if it is taken as instructed.
Time Frame: During the BPS (mean duration of approximately 3-4 weeks)
Population: Participants in the full analysis set with observations
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo SLIT-tablet | Tree SLIT-tablet
Number analyzed (Participants) | 167 | 161
score on a scale | 0.98 (0.09) | 0.97 (0.09)
Statistical Analysis 1: Comparison: Placebo SLIT-tablet vs Tree SLIT-tablet; Multiple imputation was used to impute missing data under the hypothetical strategy. The endpoint was analysed in each dataset in a linear mixed effects (LME) model with treatment and cohort as fixed effects, and pollen station within cohort as a random effect. Each treatment group was allowed different residual errors. Observed p-value; Test type: Superiority; p = 0.9277, Mixed Models Analysis; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.21 to 0.23] — Placebo SLIT-tablet vs tree SLIT-tablet

24. Secondary Outcome: Average Weekly Overall Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Score During the Tree Pollen Season (TPS) (12-17 Years Only)
Description: as for outcome 23
Time Frame: During the TPS (mean duration of approximately 11 weeks)
Population: Participants in the full analysis set with observations
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo SLIT-tablet | Tree SLIT-tablet
Number analyzed (Participants) | 172 | 166
score on a scale | 0.85 (0.07) | 0.86 (0.08)
Statistical Analysis 1: Comparison: Placebo SLIT-tablet vs Tree SLIT-tablet; Multiple imputation was used to impute missing data under the hypothetical strategy. The endpoint was analysed in each dataset in a linear mixed effect (LME) model with treatment and cohort as fixed effects, and pollen station within cohort as a random effect. Each treatment group was allowed different residual errors. Observed p-value; Test type: Superiority; p = 0.9643, Mixed Models Analysis; Mean Difference (Final Values) = -0.00, 95% CI 2-sided [-0.19 to 0.18] — Placebo SLIT-tablet vs tree SLIT-tablet

25. Secondary Outcome: Overall Paediatric Rhinoconjunctivitis Quality of Life Questionnaire (PRQLQ) Score During the Birch Pollen Season (BPS) (5-11 Years Only)
Description: The PRQLQ measured the paediatric rhinoconjunctivitis quality of life. The PRQLQ consisted of 23 items, each scored on a 7-point scale ranging 0-6, with higher scores indicating worse quality of life. The overall PRQLQ score was the mean of the 23 item scores.
  The primary estimand for the endpoint was the trial product estimand. The trial product estimand assesses the anticipated effect of the tree SLIT-tablet if it is taken as instructed.
Time Frame: During the BPS (mean duration of approximately 3-4 weeks)
Population: Participants in the full analysis set with observations
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo SLIT-tablet | Tree SLIT-tablet
Number analyzed (Participants) | 260 | 257
score on a scale | 1.30 (0.07) | 1.12 (0.07)
Statistical Analysis 1: Comparison: Placebo SLIT-tablet vs Tree SLIT-tablet; [analysis description as in outcome 24, analysis 1]; Test type: Superiority; p = 0.0287, Mixed Models Analysis; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [0.02 to 0.34] — Placebo SLIT-tablet vs. tree SLIT-tablet

26. Secondary Outcome: Treatment Satisfaction (TSQM-9)
Description: Treatment satisfaction was measured using the 9-item treatment satisfaction questionnaire for medication (TSQM-9 questionnaire). After ending treatment, participants completed the TSQM-9 questionnaire which consisted of 9 items covering 3 domains. Each item was scored on a 5 point (ranging 1-5) or 7 point (ranging 1-7) scale. For each domain, item scores were summed and normalised to a 0-100 scale, with higher scores indicating better satisfaction.
Time Frame: After ending treatment (after approximately 52 weeks of treatment)
Population: Patient-reported outcomes were collected from 479 placebo and 473 tree SLIT-tablet participants. Not all participants provided data for the 3 categories (convenience, effectiveness, and global satisfaction) resulting in different participant numbers analyzed in each category. The endpoint comprises the 3 categories, and thus to report the endpoint as one, the categories are reported together.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo SLIT-tablet | Tree SLIT-tablet
Number analyzed (Participants) | 479 | 473
score on a scale
  Convenience: number analyzed (Participants) | 459 | 456
  Convenience | 79.6 (14.7) | 78.2 (15.3)
  Effectiveness: number analyzed (Participants) | 459 | 455
  Effectiveness | 59.8 (21.1) | 67.6 (18.4)
  Global satisfaction: number analyzed (Participants) | 459 | 455
  Global satisfaction | 62.1 (23.5) | 69.9 (20.0)

27. Secondary Outcome: Patient-rated Global Evaluation of Treatment Efficacy
Description: The global evaluation measured patient treatment satisfaction. After ending treatment, participants were asked: 'Compared to your rhinitis and/or conjunctivitis symptoms in the previous birch/tree pollen season, how have you felt overall in this birch/tree pollen season?'. The endpoint was evaluated as a binary endpoint; answer options 'much better' and 'better' were categorised as improved (taking value 1), while answer options 'the same', 'worse', and 'much worse' were categorised as not improved (taking value 0).
  The primary estimand for the endpoint was he trial product estimand. The trial product estimand assesses the anticipated effect of the tree SLIT-tablet if it is taken as instructed.
Time Frame: End of treatment (after approximately 52 weeks of treatment)
Population: Participants in the full analysis set with observations
Measure: Number (95% Confidence Interval); unit: Proportion
Arm/Group | Placebo SLIT-tablet | Tree SLIT-tablet
Number analyzed (Participants) | 455 | 443
Proportion | 0.70 [0.65 to 0.74] | 0.85 [0.81 to 0.88]
Statistical Analysis 1: Comparison: Placebo SLIT-tablet vs Tree SLIT-tablet; Multiple imputation was used to impute missing data under the hypothetical strategy. The odds of having an improved treatment efficacy according to patient-rated global evaluation was analysed using a generalised linear mixed model with a logit link function. The model includes patient-rated global evaluation of treatment efficacy (improvement/no improvement) as the response variable and treatment, cohort and age group as fixed effects and pollen station as random effects. Observed p-value; Test type: Superiority; p < 0.0001, Generalized linear mixed model (GLMM); Odds Ratio (OR) = 0.42, 95% CI 2-sided [0.30 to 0.58] — Odds ratio is (odds placebo SLIT-tablet/ odds tree SLIT-tablet)

28. Secondary Outcome: Change From Baseline in Birch Specific IgE
Description: Birch specific IgE reflects the allergen-specific allergy immunotherapy-induced immune modulation
Time Frame: From baseline (screening) to visit 4 (pre-TPS) (after approximately 19 weeks of treatment, on average) and from baseline (screening) to visit 6 (end of treatment) (after approximately 44 weeks of treatment, on average)
Population: Birch specific IgE levels were measured in 479 placebo and 473 tree SLIT-tablet participants. Data were not provided by all participants for both visit 4 and visit 6, thus the overall number of participants analyzed differs from the number analyzed at the specified visits.
Measure: Mean (95% Confidence Interval); unit: Log10 transformed kU/L
Arm/Group | Placebo SLIT-tablet | Tree SLIT-tablet
Number analyzed (Participants) | 479 | 473
Log10 transformed kU/L
  Birch specific IgE, visit 4: number analyzed (Participants) | 454 | 449
  Birch specific IgE, visit 4 | -0.21 [-0.24 to -0.18] | 0.22 [0.18 to 0.26]
  Birch specific IgE, visit 6: number analyzed (Participants) | 448 | 445
  Birch specific IgE, visit 6 | 0.10 [0.07 to 0.13] | 0.06 [0.02 to 0.10]
Statistical Analysis 1: Comparison: Placebo SLIT-tablet vs Tree SLIT-tablet; Change from baseline (screening) to visit 4 (pre-TPS). Change from baseline of log transformed concentrations is analyzed in a mixed effects linear model including treatment, visit, and treatment-visit-interaction as fixed effects, log(baseline concentration) as a covariate and subject as random effect. Observed p-value; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.43, 95% CI 2-sided [0.38 to 0.48] — Tree SLIT-tablet vs placebo SLIT-tablet, visit 4
Statistical Analysis 2: Comparison: Placebo SLIT-tablet vs Tree SLIT-tablet; Change from baseline (screening) to visit 6 (end of treatment). Change from baseline of log transformed concentrations is analysed in a mixed effects linear model including treatment, visit, and treatment-visit-interaction as fixed effects, log(baseline concentration) as a covariate and subject as random effect. Observed p-value; Test type: Superiority; p = 0.1038, Mixed Models Analysis; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.09 to 0.01] — Tree SLIT-tablet vs. placebo SLIT-tablet, visit 6

29. Secondary Outcome: Change From Baseline in Birch Specific IgG4
Description: Birch specific IgG4 reflects the allergen-specific allergy immunotherapy-induced immune modulation.
Time Frame: as for outcome 28
Population: Birch specific IgG4 levels were measured in 479 placebo and 473 tree SLIT-tablet participants. Data were not provided by all participants for both visit 4 and visit 6, thus the overall number of participants analyzed differs from the number analyzed at the specified visits.
Measure: Mean (95% Confidence Interval); unit: Log10 transformed mg/L
Arm/Group | Placebo SLIT-tablet | Tree SLIT-tablet
Number analyzed (Participants) | 479 | 473
Log10 transformed mg/L
  Birch specific IgG4, visit 4: number analyzed (Participants) | 454 | 449
  Birch specific IgG4, visit 4 | -0.09 [-0.11 to -0.07] | 0.43 [0.39 to 0.47]
  Birch specific IgG4, visit 6: number analyzed (Participants) | 448 | 445
  Birch specific IgG4, visit 6 | 0.05 [0.03 to 0.07] | 0.54 [0.51 to 0.58]
Statistical Analysis 1: Comparison: Placebo SLIT-tablet vs Tree SLIT-tablet; Change from baseline (screening) to visit 4 (pre-TPS). Change from baseline of log transformed concentrations is analysed in a mixed effects linear model including treatment, visit, and treatment-visit-interaction as fixed effects, log(baseline concentration) as a covariate and subject as random effect. Observed p-value; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.53, 95% CI 2-sided [0.48 to 0.57] — Tree SLIT-tablet vs. placebo SLIT-tablet, visit 4
Statistical Analysis 2: Comparison: Placebo SLIT-tablet vs Tree SLIT-tablet; [analysis description as in outcome 28, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.49, 95% CI 2-sided [0.45 to 0.53] — Tree SLIT-tablet vs placebo SLIT-tablet, visit 6

30. Secondary Outcome: Change From Baseline in Birch Specific IgE-Blocking Factor (IgE-BF)
Description: The IgE-blocking factor assesses the effect of serum components (including IgE-blocking antibodies known to be induced by allergy immunotherapy) competing with IgE for binding to allergen. IgE-blocking factor is calculated as 1-(S/T), where S is the amount of allergen-specific IgE bound to allergen in the (possible) presence of competing components, and where T is the total amount of allergen-specific IgE capable of binding to allergen when all competing antibodies/components have been washed off. IgE-blocking factor values closer to 0 indicate the presence of fewer IgE-blocking components and values closer to 1 indicate that more IgE is blocked from binding to the allergen.
Time Frame: as for outcome 28
Population: Birch specific IgE-BF levels were measured in 132 placebo and 119 tree SLIT-tablet participants. Data were not provided by all participants for both visit 4 and visit 6, thus the overall number of participants analyzed differs from the number analyzed at the specified visits.
Measure: Mean (95% Confidence Interval); unit: Unitless
Arm/Group | Placebo SLIT-tablet | Tree SLIT-tablet
Number analyzed (Participants) | 132 | 119
Unitless
  Birch specific IgE-BF, visit 4: number analyzed (Participants) | 127 | 113
  Birch specific IgE-BF, visit 4 | -0.01 [-0.03 to 0.01] | 0.28 [0.23 to 0.32]
  Birch specific IgE-BF, visit 6: number analyzed (Participants) | 107 | 92
  Birch specific IgE-BF, visit 6 | 0.04 [0.02 to 0.05] | 0.35 [0.30 to 0.40]
Statistical Analysis 1: Comparison: Placebo SLIT-tablet vs Tree SLIT-tablet; [analysis description as in outcome 28, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.29, 95% CI 2-sided [0.24 to 0.33] — Tree SLIT-tablet vs. placebo SLIT-tablet, visit 4
Statistical Analysis 2: Comparison: Placebo SLIT-tablet vs Tree SLIT-tablet; [analysis description as in outcome 28, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 0.31, 95% CI 2-sided [0.26 to 0.36] — Tree SLIT-tablet vs. placebo SLIT-tablet, visit 6

31. Secondary Outcome: Change From Baseline in Alder, Hazel and Oak Specific IgE
Description: Change in alder, hazel and oak specific IgE reflects the allergen-specific allergy immunotherapy-induced immune modulation.
Time Frame: as for outcome 28
Population: Alder, hazel and oak specific IgE levels were measured in 132 placebo and 119 tree SLIT-tablet participants. Data were not provided by all participants for both visit 4 and visit 6, thus the overall number of participants analyzed differs from the number analyzed at the specified visits.
Measure: Mean (Standard Deviation); unit: log10 transformed kU/L
Arm/Group | Placebo SLIT-tablet | Tree SLIT-tablet
Number analyzed (Participants) | 132 | 119
log10 transformed kU/L
  Alder specific IgE, visit 4: number analyzed (Participants) | 128 | 117
  Alder specific IgE, visit 4 | -0.22 (0.20) | 0.17 (0.41)
  Alder specific IgE, visit 6: number analyzed (Participants) | 109 | 95
  Alder specific IgE, visit 6 | 0.18 (0.34) | 0.10 (0.31)
  Hazel specific IgE, visit 4: number analyzed (Participants) | 128 | 117
  Hazel specific IgE, visit 4 | -0.22 (0.21) | 0.15 (0.38)
  Hazel specific IgE, visit 6: number analyzed (Participants) | 109 | 95
  Hazel specific IgE, visit 6 | 0.20 (0.36) | 0.11 (0.30)
  Oak specific IgE, visit 4: number analyzed (Participants) | 128 | 117
  Oak specific IgE, visit 4 | -0.21 (0.17) | 0.14 (0.37)
  Oak specific IgE, visit 6: number analyzed (Participants) | 109 | 95
  Oak specific IgE, visit 6 | 0.20 (0.34) | 0.11 (0.29)

32. Secondary Outcome: Change From Baseline in Alder, Hazel and Oak Specific IgG4
Description: Change in alder, hazel and oak specific IgG4 reflects the allergen-specific allergy immunotherapy-induced immune modulation.
Time Frame: as for outcome 28
Population: Alder, hazel and oak specific IgG4 levels were measured in 132 placebo and 119 tree SLIT-tablet participants. Data were not provided by all participants for both visit 4 and visit 6, thus the overall number of participants analyzed differs from the number analyzed at the specified visits.
Measure: Mean (Standard Deviation); unit: log10 transformed mg/L
Arm/Group | Placebo SLIT-tablet | Tree SLIT-tablet
Number analyzed (Participants) | 132 | 119
log10 transformed mg/L
  Alder specific IgG4, visit 4: number analyzed (Participants) | 128 | 117
  Alder specific IgG4, visit 4 | -0.08 (0.18) | 0.38 (0.39)
  Alder specific IgG4, visit 6: number analyzed (Participants) | 109 | 95
  Alder specific IgG4, visit 6 | 0.13 (0.26) | 0.51 (0.41)
  Hazel specific IgG4, visit 4: number analyzed (Participants) | 128 | 117
  Hazel specific IgG4, visit 4 | -0.08 (0.19) | 0.35 (0.39)
  Hazel specific IgG4, visit 6: number analyzed (Participants) | 109 | 95
  Hazel specific IgG4, visit 6 | 0.11 (0.24) | 0.46 (0.42)
  Oak specific IgG4, visit 4: number analyzed (Participants) | 128 | 117
  Oak specific IgG4, visit 4 | -0.07 (0.14) | 0.28 (0.39)
  Oak specific IgG4, visit 6: number analyzed (Participants) | 109 | 95
  Oak specific IgG4, visit 6 | 0.08 (0.21) | 0.32 (0.35)

33. Secondary Outcome: Change From Baseline in Alder and Hazel Specific IgE- Blocking Factor (IgE-BF)
Description: as for outcome 30
Time Frame: From baseline (screening) to visit 4 (pre-TPS) (after approximately 19 weeks of treatment, on average) and from baseline (screening) to visit 6 (end of treatment) (after approximately 44 weeks treatment, on average)
Population: Alder and hazel specific IgE-BF levels were measured in 132 placebo and 119 tree SLIT-tablet participants. Data were not provided by all participants for both visit 4 and visit 6, thus the overall number of participants analyzed differs from the number analyzed at the specified visits.
Measure: Mean (Standard Deviation); unit: Unitless
Arm/Group | Placebo SLIT-tablet | Tree SLIT-tablet
Number analyzed (Participants) | 132 | 119
Unitless
  Alder specific IgE-BF, visit 4: number analyzed (Participants) | 124 | 107
  Alder specific IgE-BF, visit 4 | -0.03 (0.08) | 0.20 (0.18)
  Alder specific IgE-BF, visit 6: number analyzed (Participants) | 107 | 86
  Alder specific IgE-BF, visit 6 | 0.04 (0.13) | 0.21 (0.19)
  Hazel specific IgE-BF, visit 4: number analyzed (Participants) | 118 | 104
  Hazel specific IgE-BF, visit 4 | -0.03 (0.08) | 0.15 (0.18)
  Hazel specific IgE-BF, visit 6: number analyzed (Participants) | 104 | 83
  Hazel specific IgE-BF, visit 6 | 0.02 (0.10) | 0.14 (0.17)

ADVERSE EVENTS:
Time Frame: All AEs with start date/time on or after the time of first IMP administration and no later than 7 days after last IMP administration (up to approximately 12 months).
Description: All AEs with start date/time on or after the time of first IMP administration and no later than 7 days after last IMP administration are presented including "all-cause mortality"," serious adverse events" and "other (not including serious) adverse events". Both treatment-related and non-treatment-related AEs are displayed.
Arm/Group | Placebo SLIT-tablet | Tree SLIT-tablet
All-Cause Mortality (participants affected / at risk) | 0/479 | 0/473
Serious Adverse Events (participants affected / at risk) | 6/479 | 5/473
Other Adverse Events (participants affected / at risk) | 194/479 | 315/473
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo SLIT-tablet (N=479) | Tree SLIT-tablet (N=473)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 0 (0) | 1 (1)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Lymph node abscess (Infections and infestations) | 1 (1) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Foot operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo SLIT-tablet (N=479) | Tree SLIT-tablet (N=473)
Oral pruritus (Gastrointestinal disorders) | 17 (19) | 114 (136)
Tongue pruritus (Gastrointestinal disorders) | 6 (6) | 60 (76)
Paraesthesia oral (Gastrointestinal disorders) | 8 (8) | 28 (34)
Nasopharyngitis (Infections and infestations) | 82 (124) | 81 (109)
Upper respiratory tract infection (Infections and infestations) | 43 (55) | 42 (53)
Pharyngitis (Infections and infestations) | 21 (23) | 32 (35)
COVID-19 (Infections and infestations) | 43 (44) | 27 (28)
Influenza (Infections and infestations) | 25 (27) | 17 (18)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 18 (19) | 112 (140)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication can be made before the first multi-center publication. PI shall allow Sponsor (S) not less than 60 days to review publications and 30 days to review presentations. S can comment and require removal of confidential information. Upon S request, PI must delay the publication or presentation for 6 months to permit S to file a patent application or take other steps to protect S' information. Any other public statements regarding the trial requires prior written consent from S.

DOCUMENTS (2):
  • Study Protocol (2022-05-24): https://cdn.clinicaltrials.gov/large-docs/54/NCT04878354/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-19): https://cdn.clinicaltrials.gov/large-docs/54/NCT04878354/SAP_001.pdf